CLINICAL TRIAL: NCT06074315
Title: Evaluation of the Effectiveness of Nail Genesis DLSO Product for Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nail Genesis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT002-02
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Distal Lateral Subungual Onychomycosis; Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, randomized, parallel-group, double-blind, vehicle- controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nail Genesis DLSO Product (Experimental): Nail Genesis DLSO Product, poly(urea-urethane) in carrier solvents, applied topically, once daily, to target toenail.
  Interventions: Device: Nail Genesis DLSO Product
- Vehicle (Placebo Comparator): poly(urea-urethane) in carrier solvents, applied topically, once daily, to target toenail.
  Interventions: Device: Nail Genesis DLSO Product (vehicle only)

INTERVENTIONS:
Device: Nail Genesis DLSO Product — Nail fungus is difficult to treat with topical drugs because of the thickness of the nails (Murdan, 2002). Nail Genesis DLSO Product does not contain a drug or antifungal agent and so is not designed to have a direct action on the microorganism, but instead will act by changing the conditions that allow growth of the fungus (i.e., keeping the nail plate and underlying nail bed dry and inhibiting secondary infection).
  Arms: Nail Genesis DLSO Product
Device: Nail Genesis DLSO Product (vehicle only) — The Nail Genesis DLSO product poly-urethane vehicle
  Arms: Vehicle

SUMMARY:
This is a Pre-IDE, prospective, multicenter, randomized, parallel-group, double-blind, vehicle- controlled study to evaluate safety and effectiveness of Nail Genesis DLSO Product for the treatment of DLSO compared with vehicle in infected great toenails in a total of 338 males and non-pregnant, non-lactating, females between 18 and 65 years of age (inclusive). Subjects will be randomized in a 2:1 ratio to receive either Nail Genesis DLSO Product or vehicle.

Subject eligibility will be determined during a Screening assessment. Subjects will complete a 4week washout period after discontinuation of a topical product or a 12-month washout period after discontinuation of an oral product or light-based therapy prior to randomization. Eligible subjects will be randomized in a 2:1 ratio to receive Nail Genesis DLSO Product or vehicle, respectively. During the 52-week trial, study medication will be administered once daily to the target toenail for 48 weeks.

A subject will be considered to have completed the study when he or she has completed the study assessments at Week 52. The 52-week visit is for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, and 18 to 65 years of age, inclusive.
* Subject has nail fungal infection of at least one great toenail (per visual assessment, positive KOH preparation, and positive dermatophyte culture).
* Subject has target toenail showing 20-50% involvement without matrix (lunula) involvement.
* Subject has 3 mm of unaffected nail (from proximal nail fold) on target toenail.
* Subject has target toenail thickness of 3 mm or less.
* Subject must be physically able to reach toes to clean, trim, and apply product to the target toenail.
* Subject is willing and available to return for study follow up.
* Subject or legal representative is able to understand and provide signed consent for participating in the study.
* Female subject of childbearing potential has negative urine pregnancy test.
* Females must be post-menopausal or must agree to use approved contraceptives (actions, de- vices or medications to prevent or reduce the likelihood of pregnancy) throughout the study (abstinence is NOT an accepted form of contraception).

Exclusion Criteria:

* Subject has known hypersensitivity or allergy to the product materials.
* Subject has negative KOH preparation or dermatophyte culture.
* Subject has dermatophytoma on target toenail.
* Subject is enrolled in another investigational drug, device, or product protocol that would interfere with this study.
* Subject is using other topical or pharmaceutical treatments for any nail conditions; a wash-out period of at least four weeks after discontinuation of a topical product or 12 months after discontinuation of an oral product or light-based therapy for treatment of nail fungus is required.
* Subject has history of immunosuppression and/or clinical signs indicative of possible immunosuppression.
* Subject with possible chronic disease, including: diabetes, psoriasis, immune deficiency (HIV), severe foot injury, chronic vascular disease, or in which delayed treatment (approved treatment) of DLSO for one year could present a significant health concern.
* Subject has presence of toenail infection other than dermatophytes on target toenail.
* Subject has any disease/condition that might cause toenail abnormalities or interfere with evaluation.
* Subject has had previous toenail surgery on target toenail.
* Subject is a pregnant or nursing female.
* Subject is an Investigator, Nail Genesis' personnel, or Nail Genesis' Scientific Advisory Board (SAB) members, or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness - Complete Cure | Week 48
  Proportion of subjects with Complete Cure (0% involvement of the target toenail in addition to Mycologic Cure (defined as both negative KOH stain and negative dermatophyte culture).
Safety - Adverse Events | Week 48
  Proportion of subjects with treatment-emergent AEs of Nail Genesis DLSO Product compared with vehicle control)

SECONDARY OUTCOMES:
Almost complete cure | Week 48
  Proportion of subjects achieving almost Complete Cure (< 10% clinical involvement of the target toenail) in addition to Mycologic Cure.
Mycological Cure | Week 48
  Proportion of subjects achieving Mycologic Cure of the target toenail at Week 48

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Clinical Trials Institute of Northwest Arkansas, Fayetteville, Arkansas
  - Catalina Research Institute, LLC, Montclair, California
  - Northern California Research, Sacramento, California
  - Metro Clinical Trials, San Bernardino, California
  - Doctors Research Network, South Miami, Florida
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Rochester Clinical Research, LLC, Rochester, New York
  - DermResearch, Austin, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Undecided